CLINICAL TRIAL: NCT01198457
Title: BONA (Adherence of Patients to Bonefos Therapy). Prospective Observational Non-interventional Study of Adherence of Patients to Bonefos Medication in Relation to Analgesic Effect and Incidence of Skeletal Events
Brief Title: Study to Investigate Adherence of Patients to Clodronate (Bonefos) Treatment
Acronym: BONA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 14561; BO0910CZ (Other: Company Internal)
Record Dates: First submitted 2010-07-29; First posted 2010-09-10 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Breast Neoplasms; Prostatic Neoplasms; Multiple Myeloma; Osteolysis
Keywords: Clodronate; Compliance
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Multiple Myeloma; Osteolysis; Patient Compliance | interventions — Clodronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Clodronate (Bonefos, BAY94-8393)

INTERVENTIONS:
Drug: Clodronate (Bonefos, BAY94-8393) — Random group of patients in oncology clinic

SUMMARY:
Adherence (or compliance with) a medication regimen is generally defined as the extent to which patients take medication as prescribed by their health care providers. The adherence to medications has close relation to effectiveness of the therapy. The primary objective of this study is to observe the adherence to treatment with oral clodronate (PDC, proportion of days covered, number of days in which clodronate is taken according to treating physician recommendation) in patients with malignancy. The secondary "hypothesis generating" objective is to describe the relation between adherence to treatment with oral clodronate and efficacy of the therapy (skeletal events, pain).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer, prostate cancer, multiple myeloma and other skeletal events causing tumors
* Bone metastases
* Therapy with clodronate (1600 mg per day, 800 mg tablets) according to SmPC (Summary of Product Characteristics) Bonefos.
* By agreeing to usage of patients diaries and goodwill with accounting of tablets

Exclusion Criteria:

* According to SmPC (Summary of Product Characteristics) Bonefos.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Random group of patients in oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment with oral clodronate (PDC, proportion of days covered). | 12 months of therapy.

SECONDARY OUTCOMES:
Efficacy evaluation of the therapy based on incidence of skeletal events | 12 months
Efficacy of the therapy in pain releif will be investigated exploratory based on questionnaire | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Czechia